CLINICAL TRIAL: NCT00301756
Title: A Phase 2 Study of PXD101 in Platinum Resistant Epithelial Ovarian Tumors and Micropapillary/Borderline (LMP) Ovarian Tumors
Brief Title: Belinostat in Treating Patients With Advanced Ovarian Epithelial Cancer, Primary Peritoneal Cancer, or Fallopian Tube Cancer or Ovarian Low Malignant Potential Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00144; NCI-2009-00144 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PMH-PHL-041; CDR0000459798; NCI-7267; PHL-041 (Other: University Health Network Princess Margaret Cancer Center P2C); 7267 (Other: CTEP); N01CM17107 (NIH); N01CM62203 (NIH)
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2016-12-14 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Fallopian Tube Carcinoma; Primary Peritoneal Carcinoma; Recurrent Borderline Ovarian Surface Epithelial-Stromal Tumor; Recurrent Ovarian Carcinoma; Stage III Borderline Ovarian Surface Epithelial-Stromal Tumor; Stage III Ovarian Cancer; Stage IV Borderline Ovarian Surface Epithelial-Stromal Tumor; Stage IV Ovarian Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — belinostat

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Belinostat; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Belinostat — Given IV
  Other Names: Beleodaq; PXD 101; PXD101
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well belinostat works in treating patients with ovarian epithelial cancer, primary peritoneal cancer, or fallopian tube cancer that have spread to other places in the body or ovarian low malignant potential tumors. Belinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the antitumor activity of PXD 101 as a single agent in the following patient population using objective response rates (complete and partial): a) Platinum resistant ovarian carcinoma (progression within 6 months of platinum based therapy); b) Micropapillary / borderline (Low Malignant potential) ovarian carcinoma.

SECONDARY OBJECTIVES:

I. To determine the antitumor activity of PXD 101 with regards to stable disease rates, duration of response, progression- free, median and overall survival rates as well as determine the safety and tolerability this drug.

TERTIARY OBJECTIVES:

I. To determine the relationship between clinical and pharmacodynamic effects of PXD101 in patients with platinum resistant and micropapillary tumors undergoing treatment with this drug.

OUTLINE:

Patients receive belinostat intravenously (IV) over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed ovarian epithelial cancer, primary peritoneal carcinoma or fallopian tube cancer that recurred despite initial platinumbased therapy OR micropapillary/borderline (Low Malignant Potential) tumors of ovary
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Patients in the platinum resistant (progression within 6 months of platinum based therapy) group: must have had no more than a total of 3 prior chemotherapy regimens; at least one prior regimen will have contained a platinum agent (carboplatin or cisplatin)
* Patients with micropapillary or borderline (LMP) tumors: must have had no more than a total of 3 prior chemotherapy regimens
* Patients must have completed any prior chemotherapy, radiotherapy or surgery at least 4 weeks (at least 6 weeks for nitrosureas and mitomycin C) before study entry and patients must have recovered from the toxic effects from any prior therapy; patients must not have had more than 40% of their bone marrow radiated and must have either measurable disease outside the field or progression post radiation therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Leukocytes >= 3.0 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin =< institutional upper limit of normal
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/ alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Biopsies are not mandatory but patients will be asked to undergo tumor biopsy once before and once during experimental therapy if considered medically safe for them to do so; patients must be willing to have the peripheral blood mononuclear cell (PBMC) procured prior to and during the treatment
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of PXD101 will be determined following review of their case by the Principal Investigator; efforts should be made to switch patients who are taking enzyme-inducing anticonvulsant agents to other medications
* Women of child-bearing potential and their partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* A marked baseline prolongation of QT/corrected QT (QTc) interval, e.g., repeated demonstration of a QTc interval > 500msec; long QT syndrome; the required use of concomitant medication on PXD101 infusion days that may cause Torsade de Pointes (disopyramide, dofetilide, ibutilide, procainamide, quinidine, sotalol, bepridil, amiodarone, arsenic trioxide, cisapride, lidoflazine, clarithromycin, erythromycin, halofantrine, pentamidine, sparfloxacin, domperidone, droperidol, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide & methadone)
* Significant cardiovascular disease including unstable angina pectoris, uncontrolled hypertension, congestive heart failure related to primary cardiac disease, a condition requiring anti-arrythmic therapy, ischemic or severe valvular heart disease, or a myocardial infarction within 6 months prior to the trial entry
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to sulfonamides, arginine and compounds of similar chemical or biologic composition to PXD101
* Patients should not have taken valproic acid, another histone deacytelase inhibitor, for at least 2 weeks prior to enrollment
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with bowel obstruction would not be eligible because of compromised functional status unless they are on parenteral support
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with PXD101
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-09; Primary Completion 2009-08 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Principal Investigator — University Health Network Princess Margaret Cancer Center P2C
Locations (4):
- Canada (4):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network Princess Margaret Cancer Center P2C, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Belinostat / Enzyme Inhibitor Therapy): Patients receive belinostat IV over 30 minutes on days 1-5. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Belinostat / Enzyme Inhibitor Therapy)
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 6
Age, Continuous [Median (Full Range); unit: years] | 54 [28 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Region of Enrollment [Number; unit: participants]
  Canada | 32

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Belinostat in Terms of Complete or Partial Response; Disappearance of All Target Lesions or at Least a 30% Decrease in the Sum of the Longest Diameter of Target Lesions, Taking as Reference the Baseline Sum LD
Description: Efficacy of belinostat in terms of complete or partial response; disappearance of all target lesions or at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) or Rustin criteria.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 32
participants | 0

2. Secondary Outcome: Time to Disease Progression (Epithelial Ovarian Cancer Group)
Description: Assessed by RECIST criteria. Summarized using summary statistics, such as the mean, median, counts and proportion.
Time Frame: Up to 5 years
Population: Eighteen patients with Epethelial Ovarian Cancer were analyzed
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
months | 2.3 [1.2 to 5.7]

3. Secondary Outcome: Stable Disease Rate, Defined as Neither Sufficient Shrinkage to Qualify for PR Nor Sufficient Increase to Qualify for PD, Taking as Reference the Smallest Sum LD Since the Treatment Started (Low Malignant Potential Group)
Description: Stable disease rate, defined as neither sufficient shrinkage to qualify for Partial Response nor sufficient increase to qualify for Progressive disease, taking as reference the smallest sum LD since the treatment started. Summarized using summary statistics, such as the mean, median, counts and proportion. Assessed by RECIST criteria.
Time Frame: Up to 5 years
Population: 14 patients with Low Malignant Potential tumours or Micropapillary / borderline were analyzed
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 14
participants | 10

4. Secondary Outcome: Duration of Response
Description: Summarized using summary statistics, such as the mean, median, counts and proportion. Ninety-five percent confidence intervals will be constructed and selected results will be illustrated using figures and plots.
Time Frame: From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 5 years
Population: No participants had an objective response out of the 32 patients analyzed.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival
Description: Computed using the Kaplan-Meier method. Ninety-five percent confidence intervals will be constructed and selected results will be illustrated using figures and plots.
Time Frame: Duration of time from start of treatment to time of progression, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 12
months | 13.4 [5.6 to NA] — 95% confidence interval, 5.6 to not reached

6. Secondary Outcome: Overall Survival
Description: as for outcome 5
Time Frame: Up to 5 years
Population: Data were not collected
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Grade 3 Adverse Events Using the National Cancer Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: Events of Thrombosis, Hypersensitivity and ALP will be tabulated.
Time Frame: Up to 5 years
Population: 18 patients with Epithelial ovarian cancer (EOC) and 14 patients with Micro-papillary ovarian tumor (LMP)
Measure: Number; unit: events
Arm/Group | Treatment (Belinostat / Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 32
events | 5

8. Secondary Outcome: Time to Disease Progression (Low Malignant Potential or Micropapillary / Borderline Ovarian Tumour Group)
Description: Assessed by RECIST criteria. Summarized using summary statistics, such as the mean, median, counts and proportion.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 14
months | 13.4 [5.6 to NA] — A value is not available because the upper range was not reached

9. Secondary Outcome: Stable Disease Rate, Defined as Neither Sufficient Shrinkage to Qualify for PR Nor Sufficient Increase to Qualify for PD, Taking as Reference the Smallest Sum LD Since the Treatment Started (Epithelial Ovarian Cancer Group)
Description: Stable disease rate, defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started. Summarized using summary statistics, such as the mean, median, counts and proportion. Assessed by RECIST criteria.
Time Frame: Up to 5 years
Population: 18 patients from Epithelian Ovarian Cancer patients were analyzed
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 18
participants | 9

10. Other Pre Specified Outcome: Relationship Between Clinical and Pharmacodynamic Effects of Belinostat in Patients With Platinum Resistant and Micropapillary/ Borderline Ovarian Tumors
Description: Summarized using summary statistics, such as the mean, median, and range. Tested using one-sample t-tests or Wilcoxon rank sum tests. Logistic regression analysis will be used to test significance.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 12/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=32)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Cytokine release syndrome (Immune system disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Hypotension (Vascular disorders) | 1
Pleural infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Activated partial thromboplastin time prolonged (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=32)
Fatigue (General disorders) | 28
Nausea (Gastrointestinal disorders) | 26
Lymphocyte count decreased (Investigations) | 24
Constipation (Gastrointestinal disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less